CLINICAL TRIAL: NCT02417116
Title: Tear Osmolarity Clinical Utility in Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Collaborators: TearLab Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP00128
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Minims Saline (Preservative Free) lubricant eye drops - daily for 90 days
  Interventions: Other: Saline
- Hypromellose - standard treatment (Active Comparator): Tear Supplement: Hypromellose 0.3% eye drops - daily for 90 days
  Interventions: Other: Tear supplement
- Combination treatment (Active Comparator): Tear Supplement 2: Hylo-Forte 0.2% Sodium Hyaluronate eye drops, Omega 3 nutrition supplement: Omega-3 tablets, Eye bag: TranquilEyes Moist Heat Lid Compresses - Daily for 90 days;
  Interventions: Other: Tear supplement 2; Dietary Supplement: Omega 3 nutrition supplement; Device: Eye bag

INTERVENTIONS:
Other: Tear supplement — Application as required to improve comfort
  Other Names: Hypermellose 0.3% eye drop
  Arms: Hypromellose - standard treatment
Other: Tear supplement 2 — Application as required to improve comfort
  Other Names: Hylo-Forte 0.2% Sodium Hyaluronate eye drop
  Arms: Combination treatment
Dietary Supplement: Omega 3 nutrition supplement — Taken each day
  Other Names: Scope Ophthalmics Omega Eye
  Arms: Combination treatment
Device: Eye bag — Applied following microwave heating to closed eyelids for 5 minutes each day
  Other Names: TranquilEyes Moist Heat Lid
  Arms: Combination treatment
Other: Saline — Application as required to improve comfort
  Other Names: Minim sodium chloride 0.9% unpreserved
  Arms: Control

SUMMARY:
Millions of people suffer from dry eye disease, causing symptoms such as redness, burning, feeling of sand or grit in the eye and light sensitivity. Dry eye disease occurs when your eyes do not produce enough tears or produce poor quality tears. This can happen for a number of reasons, including aging, hormonal changes in women and side effects of diseases or medications.

It is now possible to objectively measure the degree of dry eye disease by collecting a tiny sample of tears from the corner of the eye and then measuring the amount of salt in the tears (termed osmolarity). We aim to establish the overall levels of raised and normal tear osmolarity in people presenting to the eye clinic with complaints of dry eye, and relate this to other factors such as symptoms, topical and nutritional medication and dry eye treatment.

DETAILED DESCRIPTION:
This study will investigate the efficacy of two treatment non-pharmaceutical therapies (tear drop alone, tear drop combined with omega 3 nutritional supplement and warm compresses) for dry eye reporting patients against a control (saline) over a 3 month period. A relatively new clinical measure (osmolarity) will be performed alongside traditional tear film volume, tear film stability, gland integrity and ocular surface damage measures to determine how this influences symptomatic complaints.

ELIGIBILITY:
Inclusion Criteria:

* Dry Eye Symptoms SPEED >8

Exclusion Criteria:

* Unable to participate in 90 days therapy
* Allergic to therapy
* On medication known to affect ocular surface / tear film
* Had ocular trauma, infection or surgery
* Diagnosed with a medical condition known to affect ocular surface / tear film

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Osmolarity change | 3 months
  Salt balance in tears measured with the Tearlab

SECONDARY OUTCOMES:
Tear break-up time change | 3 months
  Tear stability following a blink
Corneal staining change | 3 months
  Fluorescein dye applied to the ocular surface and observed with blue light and a yellow filter to observe staining fluorescence
Meibomian gland change | 3 months
  Grading of meibomian glands using Oxford scale
Tear Meniscus Height | 3 months
  Height of tear meniscus along the lower lid margin observed through a slit-lamp microscope
SPEED Questionnaire change | 3 months
  Dry eye symptomology questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: James Wolffsohn, BSc MBA PhD, Principal Investigator — Aston University
Locations (6):
- United Kingdom (6):
  - Robert Frith Opticians, Shaftesbury, Dorest
  - Robert Frith Opticians, Blandford Forum, Dorset
  - Robert Frith Opticians, Gillingham, Dorset
  - Robert Frith Opticians, Twickenham, Middlesex
  - Black & Lizars Optometrists, Ayr
  - Black & Lizars Optometrists, Glasgow